CLINICAL TRIAL: NCT01136707
Title: Predictors of Adherence to Orencia
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Other Study IDs: IM101-266
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with rheumatoid arthritis new to Orencia

SUMMARY:
The purpose of this study is to examine the relationship between loading dose and adherence to Orencia.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be identified based on the presence of first infusion claim during study period for Orencia
* At least 1 medical or facility claim for rheumatoid arthritis at the time of or 6 months prior to index date
* Patients are required to be continuously enrolled for a minimum pre-index and follow-up period as detailed below
* Patients with a minimum of 3 infusion claims for Orencia
* Only those patients will be included whose first 3 infusion claims occur within 84 days

Exclusion Criteria:

* Patients less than 18 years of age at index date.
* One or more diagnoses of regional enteritis (including Crohn's disease), ulcerative colitis, anal or intestinal fistula, ankylosing spondylitis or other inflammatory spondylopathy, psoriatic arthropathy, or psoriasis any time during the 6-month pre-index period
* Patients who switch between biologics within their first three infusion claims
* Restarts, defined as those patients who go back on Orencia after a gap of 42 days
* Patients who are on other biologics at the same time as Orencia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial health plan members
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Total number of days on Orencia therapy | 6 months

SECONDARY OUTCOMES:
Rheumatoid arthritis-related and total healthcare costs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm